CLINICAL TRIAL: NCT04491136
Title: A Multicenter, Interventional, Open-label and Single-arm Study to Investigate the Effect of ARNI on Ventricular Arrhythmia in HFrEF Patients With ICD or CRT-D
Brief Title: Effective Study of ARNI on Ventricular Arrhythmia in HFrEF Patients With ICD or CRT-D (RHYTHM)
Acronym: RHYTHM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696BCN04
Record Dates: First submitted 2020-06-22; First posted 2020-07-29 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: LCZ696; sacubitril/valsartan; Heart Failure; Heart failure with reduced ejection fraction; HFrEF; Ventricular arrhythmias; Implanted Device; Healthcare resource utilization
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACEI/ARB treatment for 6 months/ARNI treatment the next 6 months (Experimental): Patients received angiotensin-converting enzyme inhibitor/angiotensin receptor blockers treatment the first 6 months. The following 6 months patients received angiotensin receptor neprilysin inhibitor treatment.
  Interventions: Drug: ACEI/ARB; Drug: ARNI

INTERVENTIONS:
Drug: ACEI/ARB — Oral ACE/ARB drug according to the investigator's discretion for the first 6 months in this study
Drug: ARNI — Oral sacubitril/valsartan at the dosage of investigators discretion, whit a target dose of 200mg bid for the next 6 months of this study
  Other Names: Entresto

SUMMARY:
The purpose of this study was to generate effectiveness data of Angiotensin receptor neprilysin inhibitor (ARNI), in the Chinese Heart failure with reduced ejection fraction (HFrEF) patients with implantable cardioverted defibrillator (ICD) or Cardiac resynchronization therapy-defibrillator (CRT-D).

DETAILED DESCRIPTION:
The rationale of this study was to compare the effect of angiotensin-converting enzyme inhibitor (ACEI) / Angiotensin receptor blockers (ARB) with the effect of ARNI on ventricular arrhythmia (VA) events for HFrEF patients with ICD or CRT-D, thus a multicenter, interventional, open-label, and prospective single-arm study was considered.

ACEI/ARB was given to the patient for 6 months. After 6 months, patients using ACEI needed to undergo a 36-hr washout period (36-hr washout period was not needed for patients using ARB at month 6). Patients then received ARNI (sponsored by Novartis only for this study).

ELIGIBILITY:
Key Inclusion criteria:

1. Male or female patients ≥18 and ≤80 years of age
2. Implanted with an ICD or CRT-D within 2 weeks
3. NYHA functional class II - IV
4. LVEF ≤40% (measured by echocardiography)
5. Signed informed consent must be obtained prior to participation in the study.

Key Exclusion criteria

1. History of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes.
2. Patient received target dose (≥200 mg/d) of ARNI for 2 weeks continuously within the 6-week period prior to study enrollment.
3. Participation in other clinical studies 3 months prior to participating study.
4. Advanced cancer or other significant comorbidities with life expectancy of <1 year.
5. Previous history of angioedema associated with ACEI/ARB treatment, hereditary or idiopathic angioedema.
6. Patients with renal artery stenosis history.
7. Current stage D HF patients requiring vasoactive drugs.
8. Symptomatic hypotension < 100/60 mmHg at visit 1 (screening) or Symptomatic hypotension < 90/60 mmHg in anti-hypertension drug treatment at visit 1 (screening).
9. Serum potassium >5.4 mmol/L at visit 1 (screening).
10. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 as measured at visit 1 (screening).
11. Pregnant or nursing (lactating) women.
12. Other exclusion depend on investigator's discretion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- China (20):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 23 investigative sites in China
Pre-assignment Details: All patients provided written informed consent prior to the start of any study-related activities.
Groups:
- ACEI/ARB Followed by ARNI: Patients received angiotensin-converting enzyme inhibitor/angiotensin receptor blockers treatment the first 6 months. The following 6 months patients received angiotensin receptor neprilysin inhibitor treatment.
Period: Overall Study
Arm/Group | ACEI/ARB Followed by ARNI
Started | 201
Safety Set (SS) (all patients who received at least one dose of study treatment.) | 201
Efficacy Analysis Set (EAS) (Patients in the safety set who received at least one dose of ARNI and completed 12 months of treatment and follow-up or withdrew early after receiving at least one dose of ARNI.) | 140
Completed | 122
Not Completed | 79
Not completed — Patient withdraw informed consent | 9
Not completed — Adverse Event | 2
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 45
Not completed — sponsor terminated the study early | 16
Not completed — Patient/guardian's decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | ACEI/ARB Followed by ARNI
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 201

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Paired Patients With Ventricular Arrhythmia (VA) Events
Description: VA events were measured through devices to determine sustained ventricular tachycardia (SVT), non-sustained ventricular tachycardia (NSVT) and premature ventricular contraction (PVC).
  SVT was defined as tachycardia lasting for ≥30 seconds or with hemodynamic disorder as determined by Holter and/or device.
  NSVT was defined as recorded by Holter and/or device. PVC was defined as an early ventricular depolarization as determined by the device, and/or detected by Holter.
  PVC data were not available for patients with single -lumen implantation type
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: Efficacy analysis set (EAS): Patients in the safety set who received at least one dose of ARNI and completed 12 months of complete treatment and follow-up or withdrew early after receiving at least one dose of ARNI. Only subjects who had this measurement index successfully paired (ACEI/ARB treatment and ARNI treatment) were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- ACEI/ARB: Patients received angiotensin-converting enzyme inhibitor/angiotensin receptor blockers treatment the first 6 months.
- ARNI: The following 6 months patients received angiotensin receptor neprilysin inhibitor treatment (sacubitril/valsartan).
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 76 | 76
Participants
  At least one SVT occurred | 13 | 12
  At least one NSVT occurred: number analyzed (Participants) | 74 | 74
  At least one NSVT occurred | 23 | 21
  At least one PVC occurred: number analyzed (Participants) | 50 | 50
  At least one PVC occurred | 40 | 38
Statistical Analysis 1: Comparison: ACEI/ARB vs ARNI; At least one SVT occurred; Test type: Other; p > 0.9999, McNemar
Statistical Analysis 2: Comparison: ACEI/ARB vs ARNI; At least one NSVT occurred; Test type: Other; p = 0.7905, McNemar
Statistical Analysis 3: Comparison: ACEI/ARB vs ARNI; At least one PVC occurred; Test type: Other; p = 0.6250, McNemar

2. Secondary Outcome: Pairwise Number of SVT, NSVT, PVC, ICD or CRT-D Shocks and ATP Events Experienced by Patients
Description: To assess the number of occurrences of Ventricular arrhythmia (VA) events and Implantable cardioverter defibrillator (ICD) or Cardiac resynchronization therapy-defibrillator (CRT-D) shocks over 6 months of ACEI/ARB and 6 months of ARNI treatment.
  PVC data were not available for patients with single-lumen implantation type
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: as for outcome 1
Measure: Number; unit: number of events
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 87 | 87
number of events
  SVT: number analyzed (Participants) | 76 | 76
  SVT | 170 | 117
  NSVT: number analyzed (Participants) | 74 | 74
  NSVT | 5353 | 1648
  PVC: number analyzed (Participants) | 50 | 50
  PVC | 9676979 | 17482398
  ICD or CRT-D shock: number analyzed (Participants) | 57 | 57
  ICD or CRT-D shock | 6 | 5
  ATP | 217 | 156

3. Secondary Outcome: Left Ventricular Ejection Fraction
Description: To compare the changes in Left Ventricular Ejection Fraction (LVEF) between ACEI/ARB and ARNI treatments.
  LVEF is a measurement expressed as a percentage of how much blood in the left ventricle is pumped out with each contraction of the heart.
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: Efficacy analysis set (EAS): Patients in the safety set who received at least one dose of ARNI and completed 12 months of complete treatment and follow-up or withdrew early after receiving at least one dose of ARNI. Only participants with assessment of LVEF at 6 months of ACEI/ARB treatment and 6 months of ARNI treatment are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of ejected blood
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 108 | 108
percentage of ejected blood | 38.84 (9.923) | 41.24 (10.021)
Statistical Analysis 1: Comparison: ACEI/ARB vs ARNI; Test type: Other; p = 0.0008, Wilcoxon signed-rank; Mean Difference (Final Values) = 2.41, 95% CI 2-sided [1.11 to 3.70], Standard Error of Mean 0.653

4. Secondary Outcome: New York Heart Association Classification
Description: To compare the changes in New York Heart Association (NYHA) level between ACEI/ARB and ARNI treatments.
  NYHA classification is a subjective physician's assessment of heart failure patient's functional capacity and symptomatic status.
  Class I - No limitation of physical activity. Class II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath). Class III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV - Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: Efficacy analysis set (EAS): Patients in the safety set who received at least one dose of ARNI and completed 12 months of complete treatment and follow-up or withdrew early after receiving at least one dose of ARNI. Only participants with assessment of NYHA at 6 months of ACEI/ARB treatment and 6 months of ARNI treatment are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 109 | 109
score on a scale | 2.03 (0.499) | 2.00 (0.509)
Statistical Analysis 1: Comparison: ACEI/ARB vs ARNI; Test type: Other; p = 0.5733, Ridit analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.07 to 0.04], Standard Error of Mean 0.028

5. Secondary Outcome: N-Terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) Level
Description: To compare the changes in the N-Terminal prohormone of Brain Natriuretic Peptide(NT-proBNP) level between ACEI/ARB and ARNI treatments.
  NT-proBNP are small proteins produced in large amounts when the heart senses it needs to work harder, such as in heart failure.
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: Efficacy analysis set (EAS): Patients in the safety set who received at least one dose of ARNI and completed 12 months of complete treatment and follow-up or withdrew early after receiving at least one dose of ARNI. Only participants with assessment of NT-proBNP at 6 months of ACEI/ARB treatment and 6 months of ARNI treatment are included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 107 | 107
pg/mL | 1233.79 (1974.401) | 1002.33 (1738.400)
Statistical Analysis 1: Comparison: ACEI/ARB vs ARNI; Test type: Other; p = 0.0006, Wilcoxon signed rank test; Mean Difference (Final Values) = -231.46, 95% CI 2-sided [-415.90 to -47.02], Standard Error of Mean 93.030

6. Secondary Outcome: Number of Hospitalizations for Arrhythmia or HF Related Hospitalizations
Description: To compare the healthcare resource utilization of Heart Failure (HF) patients during ACEI/ARB and ARNI treatments
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: Efficacy analysis set (EAS): Patients in the safety set who received at least one dose of ARNI and completed 12 months of complete treatment and follow-up or withdrew early after receiving at least one dose of ARNI.
Measure: Number; unit: number of hospitalizations
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 140 | 140
number of hospitalizations
  Number of hospitalizations | 25 | 16
  Number of hospitalizations for heart failure | 13 | 3

7. Primary Outcome: Proportion of Paired Patients Who Experienced at Least One ICD or CRT-D Shock and ATP Event
Description: Once VA events were detected, implantable cardioverter defibrillator (ICD) could treat with high-energy shocks or Anti-tachycardia pacing (ATP). ATP consists of one or more trains of pacing stimuli, expressed as a percentage of the tachycardia cycle length for a given RR interval, from the onset of the preceding R wave.
  Patients with sustained VA events would receive ICD or cardiac resynchronization therapy-defibrillator (CRT-D) shock therapy.
Time Frame: Up to 12 months (6 months of ACEI/ARB treatment and 6 months of ARNI treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI/ARB | ARNI
Number analyzed (Participants) | 87 | 87
Participants
  Occurrence of at least one ICD or CRT-D shock: number analyzed (Participants) | 57 | 57
  Occurrence of at least one ICD or CRT-D shock | 3 | 2
  Occurrence of at least one ATP event | 15 | 8
Statistical Analysis 1: Comparison: ACEI/ARB vs ARNI; Occurrence of at least one shock; Test type: Other; p > 0.9999, McNemar
Statistical Analysis 2: Comparison: ACEI/ARB vs ARNI; Occurrence of at least one ATP event; Test type: Other; p = 0.0654, McNemar

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment. Patients were followed up for 6 months for each treatment, up to a maximum duration of 13 months
Groups:
- ARNI: The following 6 months patients received angiotensin receptor neprilysin inhibitor treatment
Arm/Group | ACEI/ARB | ARNI
All-Cause Mortality (participants affected / at risk) | 3/201 | 0/140
Serious Adverse Events (participants affected / at risk) | 38/201 | 19/140
Other Adverse Events (participants affected / at risk) | 99/201 | 58/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACEI/ARB (N=201) | ARNI (N=140)
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arrhythmic storm (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 15 | 4
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 4 | 2
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Complication associated with device (General disorders) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Lead dislodgement (Product Issues) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACEI/ARB (N=201) | ARNI (N=140)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Red blood cell abnormality (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Cardiac dysfunction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 2
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular pre-excitation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 4 | 0
Chest discomfort (General disorders) | 5 | 4
Chest pain (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 3 | 0
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Immunodeficiency (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 1 | 1
Eye infection (Infections and infestations) | 0 | 1
Laryngopharyngitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 3
Urinary tract infection (Infections and infestations) | 1 | 1
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in throat (Injury, poisoning and procedural complications) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood bilirubin unconjugated increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose abnormal (Investigations) | 0 | 4
Blood glucose decreased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 1 | 1
Blood pressure decreased (Investigations) | 3 | 0
Blood urea increased (Investigations) | 0 | 1
Brain natriuretic peptide increased (Investigations) | 1 | 0
Coagulation test abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 2 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 1 | 0
Lipids increased (Investigations) | 0 | 3
Lipoprotein (a) increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
Urinary occult blood positive (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Sodium retention (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 11 | 2
Headache (Nervous system disorders) | 1 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 1
Poor quality sleep (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 3 | 1
Renal impairment (Renal and urinary disorders) | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 1
Hypotension (Vascular disorders) | 15 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT04491136/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT04491136/SAP_001.pdf